CLINICAL TRIAL: NCT05357664
Title: Multi-Center, Non-Controlled, Prospective Radiostereometric Analysis of the PINNACLE® Dual Mobility Construct
Brief Title: PINNACLE® DM RSA Study
Acronym: PIN DM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision made not to fund study
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSJ_2019_02
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis; Degenerative Arthritis; Revision Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Total Hip Arthroplasty (Experimental): Pinnacle acetabular shells used with PINNACLE DM Metal liner and BIMENTUM ALTRX PE liner with DePuy metal or ceramic heads and DePuy femoral prostheses
  Interventions: Device: Total Hip Arthroplasty
- Revision Total Hip Arthroplasty (Experimental): Pinnacle acetabular shells used with Pinnacle DM Metal liner and BIMENTUM ALTRX PE liner with DePuy metal or ceramic heads and DePuy femoral prostheses
  Interventions: Device: Revision Total Hip Arthroplasty

INTERVENTIONS:
Device: Total Hip Arthroplasty — Pinnacle acetabular shells used with PINNACLE DM Metal liner and BIMENTUM ALTRX PE liner with DePuy metal or ceramic heads and DePuy femoral prostheses
  Other Names: THA
  Arms: Total Hip Arthroplasty
Device: Revision Total Hip Arthroplasty — Pinnacle acetabular shells used with Pinnacle DM Metal liner and BIMENTUM ALTRX PE liner with DePuy metal or ceramic heads and DePuy femoral prostheses
  Other Names: RTHA
  Arms: Revision Total Hip Arthroplasty

SUMMARY:
The primary objective is to establish the mean superior cup migration of the PINNACLE® Dual Mobility Construct using model-based RSA over the first two years post-implantation. The primary endpoint is the mean vertical subsidence (Y translation, also known as superior cup migration) at 2 years as measured with RSA. Additionally, the data from this study will be compared to historical PINNACLE® data obtained in study DSJ_2018_02.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals requiring primary THA for:

   1. a severely painful and/or disabled joint (typically due to non-inflammatory degenerative joint disease).
   2. failed previous hip surgery.
   3. or dislocation risks.
2. Individuals who are able to speak, read and comprehend the informed patient consent document and willing and able to provide informed patient consent for participation in the study and have authorized the transfer of his/her information to DePuy Synthes.
3. Individuals who are willing and able to return for follow-up as specified by the study protocol.
4. Individuals who are a minimum age of 21 years at the time of consent.
5. Individuals who are willing and able to complete the Subject Hip Outcomes questionnaires as specified by the study protocol.

   -

Exclusion Criteria:

1. Individuals have active local or systemic infection.
2. Individuals who have loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb rendering the procedure unjustified.
3. Individuals with poor bone quality, such as osteoporosis, where in the surgeon's opinion, there could be considerable migration of the prosthesis or a significant chance of bone fracture and/or the lack of adequate bone to support the implant(s).
4. Individuals with Charcot's or Paget's disease.
5. Individuals who, in the judgement of the investigator, would not be a candidate for protocol allowable components to be used for their THA.
6. Women who are pregnant or lactating.
7. Individuals who have had a contralateral hip that was implanted less than 6 months prior to the time of consent into this study or individuals that expect to have a contralateral hip implanted in the 6 months following the time of consent into this study.
8. Individuals that have amputations in either leg that would impact rehabilitation following surgery.
9. Individuals who are bedridden per the Investigators determination
10. Individuals that have participated in a clinical investigation with an investigational product (drug or device) in the last three months.
11. Individuals currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
12. Individuals, in the opinion of the Investigator, who are drug or alcohol abusers or have a psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.
13. Individuals diagnosed and taking prescription medications to treat a muscular disorder that limits mobility due to sever stiffness and pain such as fibromyalgia or polymyalgia.
14. Subject has a medical condition with less than 2 years life expectancy.
15. Individual has a BMI >45 kg/m2.
16. Individuals who require revision arthroplasty and have a well-fixed non-DePuy Synthes femoral stem or a well-fixed DePuy Synthes femoral stem that does not have a polished neck

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — Concordia Joint Replacement Group, Concordia Hip and Knee Institute & University of Manitoba
Locations (3):
- Canada (3):
  - Concordia Joint Replacement Group, Concordia Hip and Knee Institute & University of Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre & Dalhousie University, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at https://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were selected for recruitment into the study from the general diagnosis populations defined as "primary total hip arthroplasty" (THA) and "revision total hip arthroplasty" (RTHA). The investigation was conducted at two centers.
Units Other Than Participants: Hips
Groups:
- PINNACLE Dual Mobility System: PINNACLE® Acetabular Cup, PINNACLE® CoCrMo Dual Mobility Metal Liner, a BI-MENTUM™ ALTRX® Dual Mobility Polyethylene Liner, a DePuy femoral stem with a polished femoral neck and a DePuy modular, femoral head PINNACLE® Dual Mobility Metal Liners and Porous-coated PINNACLE® Acetabular Cups are intended for cementless applications.
Period: Overall Study
Arm/Group | PINNACLE Dual Mobility System
Started (11) | 11; 11 Hips
Completed (0) | 0; 0 Hips
Not Completed | 11; 11 Hips

BASELINE CHARACTERISTICS:
Units Other Than Participants: Hips
Arm/Group | PINNACLE Dual Mobility System
Number analyzed (Participants) | 11
Number analyzed (Hips) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: A measurement was missed for one participant and BMI could not be calculated
  kg/m2
    number analyzed (Participants) | 10
    (all) | 29.4 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Superior Cup Migration
Description: Radiostereometric analysis (RSA) measured mean superior cup migration (Y translation in MM)
Time Frame: 2 years
Population: Study subjects who reach two years follow-up will undergo radiostereometric analysis of the study hip to determine if the acetabular cup has migrated from its post-operative position. Please note: data is not reported because the study was terminated at 6 weeks, therefore 2-year radiostereometric analyses could not be performed.
Units Other Than Participants: mm
Groups:
- Superior Acetabular Cup Migration: RSA measured mean superior cup migration (subsidence: Y translation in mm) at 2 years
Arm/Group | Superior Acetabular Cup Migration
Number analyzed (Participants) | 0
Number analyzed (mm) | 0

2. Secondary Outcome: Harris Hip Score
Description: The Harris Hip Score (HHS) has 10 items with four subscales comprising a minimum of 0 points and a maximum of 100 points with higher scores representing better function and outcomes. The four subscales include: pain severity, activities of daily living, absence of deformity and range of motion. Scoring is done according to the following: 90-100 = excellent, 80-89 = good, 70-79 = fair, 60-69 = poor, and below 60 is a failed result
Time Frame: 6 weeks post operative
Population: All study subjects who received a PINNACLE Dual Mobility implant will have their operative hip assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Hips
Groups:
- Harris Hip Score: All study subjects who received a PINNACLE Dual Mobility Implant were evaluated using the Harris Hip Score
Arm/Group | Harris Hip Score
Number analyzed (Participants) | 10
Number analyzed (Hips) | 10
units on a scale | 79.7 (9.63)

3. Secondary Outcome: HOOS Jr Score
Description: Hip Disability and Osteoarthritis Outcome Score, Joint Replacement (HOOS, JR) assesses patient pain (2 items), and functions of daily living (4 items). Scores range from 0 to 100 with a score of 0 indicating total hip disability and 100 indicating perfect hip health. This is a patient reported joint-specific score designed to evaluate outcomes after total hip arthroplasty
Time Frame: 6 weeks
Population: All study subjects who received a PINNACLE Dual Mobility implant were evaluated using the HOOS Jr
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Hip
Groups:
- Superior Acetabular Cup Migration: All study subjects who received a PINNACLE Dual Mobility Implant were evaluated using the HOOS Jr
Arm/Group | Superior Acetabular Cup Migration
Number analyzed (Participants) | 10
Number analyzed (Hip) | 10
Units on a scale | 75.3 (10.29)

4. Secondary Outcome: FJS-12
Description: The Forgotten Joint Score (FJS-12) is a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment. The Forgotten Joint Score consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities which suggests a better outcome
Time Frame: 6 weeks
Population: All study subjects who received a PINNACLE Dual Mobility Implant were evaluated using the FJS-12
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Hip
Groups:
- Forgotten Joint Score (FJS-12): All study subjects who received a PINNACLE Dual Mobility Implant were evaluated using the FJS-12
Arm/Group | Forgotten Joint Score (FJS-12)
Number analyzed (Participants) | 10
Number analyzed (Hip) | 10
Units on a scale | 44.4 (26)

5. Secondary Outcome: Linear Head Penetration
Description: Femoral head penetration into the polyethylene liner component will be determined and measured radiographically
Time Frame: 6 weeks, 1 year, 2 years
Population: Study subjects who received a Pinnacle Dual Mobility implant will have linear head penetration measured at specified timepoints. Please note: data is not reported because radiostereometric analyses were scheduled to be performed once all subjects had completed their visit at each interval. Since only 11 subjects were enrolled, no RSA measurements were performed prior to study closure at 6-weeks.
Units Other Than Participants: hips
Groups:
- Linear Head Penetration: RSA measured mean superior cup migration (subsidence: Y translation in mm) at 2 years
Arm/Group | Linear Head Penetration
Number analyzed (Participants) | 0
Number analyzed (hips) | 0

6. Secondary Outcome: RSA Measured Subsidence (Superior Cup Migration)
Description: Superior migration of the acetabular cup will be measured using RSA
Time Frame: 3 months, 6 months and 1 year
Population: Study subjects who received a PINNACLE Dual Mobility implant. Please note: data is not reported because radiostereometric analyses were scheduled to be performed once all subjects had completed their visit at each interval. Since only 11 subjects were enrolled, no RSA measurements were performed prior to study closure at 6-weeks.
Units Other Than Participants: Hips
Groups:
- RSA Measured Subsidence: RSA measured subsidence (superior cup migration) at 3 months, 6 months and 1 year.
Arm/Group | RSA Measured Subsidence
Number analyzed (Participants) | 0
Number analyzed (Hips) | 0

7. Secondary Outcome: Additional RSA Measurements
Description: Additional RSA measurements (X and Z translations in mm, X, Y, and Z rotations in degrees, and maximal total point motion in mm) at all time points
Time Frame: 6 weeks, 3 months, 6 months, 1 year and 2 years
Population: as for outcome 6
Units Other Than Participants: Hips
Groups:
- Additional RSA Measurements: RSA measurements (X and Z translations in mm, X, Y, and Z rotations in degrees, and maximal total point motion in mm) at all time points
Arm/Group | Additional RSA Measurements
Number analyzed (Participants) | 0
Number analyzed (Hips) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to the six-week time point
Arm/Group | PINNACLE Dual Mobility System
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 2/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PINNACLE Dual Mobility System (N=11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PINNACLE Dual Mobility System (N=11)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated prior to subjects reaching three-month timepoint; therefore, only secondary endpoint data at six-weeks was collected. RSA evaluations are performed once all subjects have completed follow-up at a protocol prescribed timepoint. Since the study was terminated following the enrollment of eleven subjects, no RSA evaluations took place.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT05357664/Prot_SAP_000.pdf